CLINICAL TRIAL: NCT06983119
Title: OPENING OF A MEMORY CLINIC IN THE PROVINCE OF PAVIA: Evaluation of Case-finding Strategies and Care for People With Cognitive Decline and Their Caregivers.
Brief Title: Case-Finding for Neurocognitive Disorders in Pavia
Acronym: C-FiND Pavia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDCD-RICORDARE_2024
Record Dates: First submitted 2025-04-14; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Dementia; Mild Cognitive Impairment
Keywords: Case-finding; Dementia; Mild Cognitive Impairment; Memory Clinic; Center for Cognitive Disorders and Dementia; Non-pharmacological intervention; Caregiver; Burden
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Detection of people reporting cognitive concerns (Other)
  Interventions: Other: Case-finding for Neurocognitive Disorders

INTERVENTIONS:
Other: Case-finding for Neurocognitive Disorders — The intervention targets individuals reporting cognitive concerns without a prior diagnosis of MCI or dementia, with participants accessing three different settings for evaluation. The first setting involves General Practitioner (GP) offices, where GPs, trained in dementia risk factors and cognitive assessment tools (such as GPcog), will identify at-risk patients and refer them for further evaluation at a Center for Cognitive Disorders and Dementia (CCDD). The second setting is the Dementia Operations Center (COD) Information Desk, a public service where neuropsychologists assess citizens who independently report cognitive disturbances. The third setting includes Open Days, public events aimed at detecting early signs of cognitive decline, where neuropsychologists will assess participants using the Addenbrooke's Cognitive Examination-III (ACE-III) and the LIBRA Index. Individuals identified as at-risk in any of the three settings will be referred for further evaluation at a CCDD.

SUMMARY:
Dementia is a global public health challenge with a heavy caregiving burden, impacting families, communities, and healthcare systems. It is a priority in healthcare planning, with focus on early diagnosis and ongoing support. This research project addresses the global public health challenge posed by dementia, focusing on early detection and comprehensive care. The research evaluates the clinical, social, and healthcare impact of two dementia-related projects in Italy:

1. the first "Ricor-Dare," aims to create an integrated network for identifying new cases of dementia or Mild Cognitive Impairment (MCI) and providing care to patients and caregivers;
2. the second involves establishing a new Center for Cognitive Disorders and Dementia (CCDD) in an area previously lacking such services.

The primary goal of this study is to assess the effectiveness of case-finding strategies promoted by the "Ricor-Dare" project for the early detection of cognitive decline. Researchers will compare three different settings in which case-finding will be conducted: at the general practitioners' offices, at the Dementia Operations Center, and at Open Days for the general population. The aim is to measure how many individuals in these three settings are diagnosed with Mild Cognitive Impairment (MCI) or dementia, compared to those identified as potential cases through cognitive testing.

The secondary goal of the study is to assess the social, care, and prevention impact of the activities offered within the two projects. This includes evaluating the experiences of patients and families who access the new CCDD in the province of Pavia, the impact of care pathways on caregivers, and comparing the effectiveness of the new CCDD with existing ones in the region of Lombardia. The study will also assess the role of the "Ricor-Dare" project in addressing the needs of patients, caregivers, and professionals, as well as the effectiveness of awareness-raising and training activities on dementia. Overall, the study aims to provide valuable insights into improving care for people with dementia and supporting their families and caregivers.

DETAILED DESCRIPTION:
Dementia is currently one of the most urgent challenges that global public health must address, with a significant caregiving burden that deeply impacts families, communities, and healthcare systems. It is a key priority in healthcare and social care planning worldwide, with growing emphasis on early diagnosis and appropriate support throughout the course of the disease. According to the World Health Organization, more than 55 million people globally have been diagnosed with dementia, and this number is expected to rise to 139 million by 2050. In Italy, approximately one million people are affected by dementia, and around 900,000 have MCI, with more than three million people directly or indirectly involved in caregiving. However, in high-income countries, the proportion of diagnosed cases remains relatively low, with estimates suggesting that only 20-50% of documented cases are diagnosed in primary care settings. The province of Pavia has 539,239 inhabitants, with an estimated 11,300 individuals diagnosed with dementia and 9,000 with MCI. Consistent with international literature, the ratio of observed to expected cases of dementia and MCI suggests a significant underestimation. Timely diagnosis of the disease or risk of disease enables the person and their caregivers to make informed choices, plan for the future, and gain access to treatments that can help manage symptoms. Centers for Cognitive Disorders and Dementia (CCDD) are healthcare services that play a critical role in the management of dementia and cognitive disorders. Scientific evidence shows that timely access to a specialized cognitive assessment and diagnostic service can lead to better outcomes for individuals with cognitive decline and their families, and be cost-effective for the healthcare system. An accurate and timely diagnosis, support for individuals with dementia and their families, along with early intervention by a multidisciplinary team of healthcare professionals, can have a positive impact on maintaining functional abilities and delaying cognitive decline and institutionalization.

The overall goal of this study is to assess the social and health impact of various services and actions aimed at individuals with cognitive decline within two projects initiated in Italy, specifically in in the Pavia area located in northern Italy: the "Ricor-Dare: integrated territorial network for dementia" project and the opening of a new Cognitive Disorders and Dementia Center (CCDD) Lomellina by Fondazione Mondino in the city of Vigevano. Specifically, the primary goal of this study is to measure the effects of case-finding strategies for the timely detection of dementia in its prodromal or early stages across three different settings. The secondary aim of this study is to evaluate and monitor the social and care effects of the activities offered within the two projects, aimed at patients, caregivers, healthcare professionals, and the community, through a series of indicators reflecting social and health care. This objective will allow for the evaluation, through a set of indicators, of the impact of these complex social and health care, and social actions both on patients identified through case-finding activities and on patients attending the new CCDD Lomellina in the province of Pavia.

For the primary goal of this study, the investigators will evaluate the impact of different case-finding strategies in identifying patients with MCI or dementia. These strategies will be implemented across three different settings:

1. General Practitioners (GPs) Offices: With their in-depth knowledge of their patients' medical histories, GPs play a crucial role in identifying those at risk of dementia or exhibiting cognitive symptoms. Using tools like the GP Cognitive Assessment of Cognition (GPcog), GPs can detect early signs of cognitive decline and refer patients for further evaluation at a CCDD. As part of the study, two annual conferences will be organized to train GPs on neurodegenerative diseases, dementia risk factors, and the GPcog. Patients scoring at the GPcog below 5 or in the borderline range (5-8) will be referred for a second-level neuropsychological evaluation at the CCDD. Additionally, a neuropsychologist will visit selected GP offices three times a year. During these visits, the neuropsychologist will conduct interviews, assess risk factors using the Lifestyle for BRAin health (LIBRA), and perform cognitive evaluations using the Addenbrooke's Cognitive Examination-III (ACE-III). Patients with below-normal or borderline ACE-III scores will be recommended for further CCDD evaluation. This initiative aims to enhance GPs' awareness of case-finding tools in their routine practice.
2. Information desk of the Dementia Operations Center (COD): The COD information desk offers a free public service aimed at the early management of citizens reporting subjective cognitive disturbances that may indicate prodromal or early-stage dementia. The case-finding strategy at the COD involves enrolling all citizens who independently report subjective cognitive disturbances without a prior diagnosis of cognitive decline. Specifically, a neuropsychologist will conduct an interview to collect demographic and medical history information, as well as dementia risk factors through the LIBRA Index, and carry out a first-level neuropsychological assessment through the ACE-III. Those scoring below the norm or borderline will be recommended for further evaluation at the CCDD.
3. Open Days: The Open Days are territorial initiatives for citizen designed for the early management of reports regarding subjective cognitive disturbances that could indicate prodromal or early-stage dementia. The case-finding strategy for Open Days involves organizing approximately two events per year, aimed at early detection of cognitive disturbances. During the Open Day, a neuropsychologist will conduct an interview to collect demographic and medical history information, as well as risk factors for dementia through the LIBRA Index, and perform a first-level neuropsychological assessment through the ACE-III. Those scoring below the norm or borderline will be recommended for further evaluation at the CCDD.

For the secondary goal of the study, the investigators will assess the experiences of patients and families who access the new CCDD in the province of Pavia, the impact of care pathways on caregivers, and comparing the effectiveness of the new CCDD with existing ones in the region of Lombardia. Below a detailed description of the six secondary outcomes are presented:

1. Explore the effect of the opening of a new CCDD. Assessing the role and contribution of the new CCDD in the management and care of individuals with dementia and MCI comparing data with other CCDDs in the Lombardy region. At the new CCDD, various diagnostic and care services are offered for patients with cognitive impairment. These include a neurological consultation to assess cognitive deterioration, followed by additional tests such as neuropsychological evaluations, neuroimaging, and advanced diagnostics at the Mondino Foundation. Multidisciplinary consultations, such as geriatrics and psychiatry, may also be recommended based on the neurologist's discretion. After the diagnostic process, patients and their families receive a joint consultation with a neurologist and psychologist to discuss the diagnosis and define a care plan. This care plan encompasses pharmacological treatments, including regular follow-ups for adjusting medications, and non-pharmacological treatments, such as individual or group cognitive stimulation. To evaluate the impact of the new CCDD's activity, data will be collected on the number of patients assessed, their diagnoses, and the services provided. An online questionnaire based on the National Survey on Cognitive Disorders and Dementia Centers will be administered to the CCDD Mondino Lomellina and Mondino Pavia to gather this data. The responses will be compared with previous survey results and regional benchmarks.
2. Explore the experience of people with cognitive decline and their caregivers accessing the new CCDD to evaluate the social and healthcare impact of opening a new CCDD. This will provide insights into challenges and needs, helping improve support throughout the diagnostic and care process. To achieve this, two methods will be employed. The first involves administering tailored questionnaires to both patients with mild dementia or MCI and their caregivers after their first follow-up visit at the CCDD. The second method includes conducting an online focus group with at least 10 caregivers, providing an opportunity to discuss their experiences with the new clinical care setup.
3. Evaluate the impact and effectiveness of diagnostic and care pathways specifically designed for caregivers, offered in the "Ricor-Dare" project and through routine clinical practice at the new CCDD. This action involves three phases: an initial evaluation (pre-test) of caregivers' burden (Zarit Burden Interview) and caregivers' preparedness to assess their perceived readiness to manage the physical and emotional needs of their loved ones (Caregiver Preparedness Scale), followed by tailored support interventions (individual psychological support, psychoeducational groups, Alzheimer's café), and a final evaluation (post-test) with the same questionnaires use in the pre-test session to assess the effectiveness of the interventions.
4. Evaluate the social and healthcare impact of the "Dementia Operations Center (COD)" as a resource for people with dementia, caregivers, and healthcare and social-care professionals. The Dementia Operations Center (COD) is the central hub of the "Ricor-Dare" project. It serves as a key point of contact for dementia-related inquiries, facilitating early intervention by directing patients, caregivers, and healthcare professionals to the appropriate services within the territorial network. The COD receives referrals from healthcare providers such as general practitioners (GPs), hospitals, nursing homes, social services, and directly from patients, caregivers, or citizens. The initial contact is made via phone, and based on an analysis of the caller's needs, further physical consultations may be recommended at the COD's information desk. With a thorough mapping of the local healthcare and social service network, COD aims to meet the needs of patients, caregivers, and professionals by providing guidance on the best path for cognitive decline management. This includes assistance with the recommended pathway, non-pharmacological treatments, and caregiver support. The COD also provides information on local healthcare services, such as CCDD, nursing homes, home care, social services, and legal processes like disability procedures. The first contact with COD is through a phone number, answered by trained psychologists or staff. If necessary, callers are referred to the physical COD desk for further evaluation.
5. Evaluate the impact of awareness and education activities on dementia. The goal is to promote social and cultural actions that improve inclusivity for people with dementia within the community. Awareness initiatives will be delivered through three annual events targeting citizens, third-sector personnel (e.g., police, firefighters), and middle and high school students.
6. Evaluate the effectiveness of training activities for healthcare and social care professionals. The objective is to assess the effectiveness of these training programs in enhancing professionals' understanding of dementia and their attitudes toward patients and caregivers. The training, provided within the Cariplo "Welfare in Aging" project - "Ricor-Dare: Integrated Territorial Dementia Network," includes annual sessions led by experts, tailored to different roles (e.g., GPs, pharmacists, nurses, healthcare assistants). To measure the training's effectiveness, participants will complete the Dementia Knowledge-20 (DK-20) and the Approaches to Dementia Questionnaire (ADQ) before (T0) and after (T1) the training. Additionally, a survey will assess the perceived utility and relevance of the training content in clinical practice.

ELIGIBILITY:
For the Primary Outcome the inclusion criteria are:

* Age 50 or older
* Assessment conducted using GPcog/ACE-III depending on the setting
* No prior diagnosis of cognitive decline
* Ability to understand the study objectives and sign an informed consent

For the Primary Outcome the exclusion criteria are:

* Age under 50
* Presence of a diagnosis of cognitive decline
* Limited knowledge of the Italian language

For the secondary outcome the inclusion criteria are:

Patient:

* All patients/people who are included in one of the actions provided through the "Ricor-Dare" Project or who are attending a visit scheduled in the clinical-care pathway of the CDCD Fondazione Mondino Pavia or Lomellina;
* Ability to understand the aims of the study and to sign an informed consent

Caregiver:

* Age equal to or greater than 18 years
* Informal caregiver of a family member with a suspected or confirmed diagnosis of dementia who is included in one of the actions provided through the "Ricor-Dare" project or who are attending a visit scheduled in the clinical-care pathway of the CDCD;
* Acceptance of informed consent and voluntary participation in the study.

Healthcare professionals:

* All healthcare and social healthcare professionals (GPs, pharmacists, nurses, nurses auxiliary) who practice in the cities of Pavia and Vigevano who participate in the project and agree to undergo assessments and training;
* Acceptance of informed consent and voluntary participation in the study.

Fo the Secondary Outcome the exclusion criteria are:

Patient:

- Inability to understand the aims of the study and to sign an informed consent

Caregiver:

* Age under 18
* Formal caregivers, i.e. any person who provides assistance to the patient in exchange for payment of a fee;
* Caregivers with limited knowledge of the Italian language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Effects of the case-finding strategy for the early detection of dementia in its prodromal or initial stages. | Up to 26 months
  The number of individuals, from the three case-finding settings, diagnosed at the CCDD with Mild Cognitive Impairment (MCI) or dementia within 26 months following assessment at case-finding compared to the total number of people identified as positive cases through GPcog and/or ACE-III and assessed within the three different case-finding settings.

SECONDARY OUTCOMES:
The impact of the new CCDD on clinical care in an area that previously lacked such services. | Up to 26 months
  Number of patients managed at the new CDCD during the study period, all of whom underwent a baseline neurological examination, a comprehensive neuropsychological assessment, and a follow-up neurological evaluation.
Patient and caregiver satisfaction with accessing the new CCDD. | Up to 26 months
  Number of completed satisfaction questionnaires from both patients and caregivers and their satisfaction regarding waiting times for the first medical appointments, satisfaction with the initial consultation, fulfillment of needs, and quality of services provided. For each item minimum score is 1 and maximum score is 5, where a higher score indicates higher satisfaction.
The impact of the diagnostic-care pathway for caregivers at CCDD and "Ricor-Dare" project. | Up to 26 months
  Number of caregivers who completed the initial and final assessments and received support interventions. The efficacy of these interventions is assessed by measuring changes in caregiver burden using the validated Zarit Burden Interview. The minimum score is 0 and the maximum score is 88, where a higher score indicates a greater caregiver burden.
The impact of the "Dementia Operations Center (COD)" pathway of the "Ricor-Dare" project. | Up to 26 months
  Number of requests received and successfully addressed through the Dementia Operations Center (COD) pathway of the 'Ricor-Dare' project.
The impact of education activities on dementia promoted by the "Ricor-Dare" project. | Up to 26 months
  Number of people reached.
Effectiveness of training activities for healthcare and social care professionals promoted by the "Ricor-Dare" project. | Up to 26 months
  Number of healthcare and social care professionals participating in the training activities. The efficacy of these training activities is assessed by measuring changes in knowledge by the validated Dementia Knowledge-20 questionnaire (DK-20). The minimum score is 0 and the maximum score is 11, where a higher score indicates a greater knowledge of dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Costa, MD, Study Director — IRCCS National Neurological Institute "C. Mondino" Foundation
Locations (1):
- IRCCS National Neurological Institute "C. Mondino" Foundation, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shanahan N, Orrell M, Schepers AK, Spector A. The development and evaluation of the DK-20: a knowledge of dementia measure. Int Psychogeriatr. 2013 Nov;25(11):1899-907. doi: 10.1017/S1041610213001142. Epub 2013 Aug 15. PMID 23947900
- [Background] Pucciarelli G, Savini S, Byun E, Simeone S, Barbaranelli C, Vela RJ, Alvaro R, Vellone E. Psychometric properties of the Caregiver Preparedness Scale in caregivers of stroke survivors. Heart Lung. 2014 Nov-Dec;43(6):555-60. doi: 10.1016/j.hrtlng.2014.08.004. Epub 2014 Sep 18. PMID 25239706
- [Background] Chattat R, Cortesi V, Izzicupo F, Del Re ML, Sgarbi C, Fabbo A, Bergonzini E. The Italian version of the Zarit Burden interview: a validation study. Int Psychogeriatr. 2011 Jun;23(5):797-805. doi: 10.1017/S1041610210002218. Epub 2010 Dec 16. PMID 21205379
- [Background] Pigliautile M, Chiesi F, Stablum F, Rossetti S, Primi C, Chiloiro D, Federici S, Mecocci P. Italian version and normative data of Addenbrooke's Cognitive Examination III. Int Psychogeriatr. 2019 Feb;31(2):241-249. doi: 10.1017/S104161021800073X. Epub 2018 Jul 19. PMID 30021668
- [Background] Franchini F, Musicco M, Ratto F, Storti G, Shofany J, Caltagirone C, Di Santo SG. The LIBRA Index in Relation to Cognitive Function, Functional Independence, and Psycho-Behavioral Symptoms in a Sample of Non-Institutionalized Seniors at Risk of Dementia. J Alzheimers Dis. 2019;72(3):717-731. doi: 10.3233/JAD-190495. PMID 31640092
- [Background] Pirani A, Brodaty H, Martini E, Zaccherini D, Neviani F, Neri M. The validation of the Italian version of the GPCOG (GPCOG-It): a contribution to cross-national implementation of a screening test for dementia in general practice. Int Psychogeriatr. 2010 Feb;22(1):82-90. doi: 10.1017/S104161020999113X. Epub 2009 Nov 6. PMID 19891815
- [Background] Banerjee S, Wittenberg R. Clinical and cost effectiveness of services for early diagnosis and intervention in dementia. Int J Geriatr Psychiatry. 2009 Jul;24(7):748-54. doi: 10.1002/gps.2191. PMID 19206079
- [Background] Steiner GZ, Ee C, Dubois S, MacMillan F, George ES, McBride KA, Karamacoska D, McDonald K, Harley A, Abramov G, Andrews-Marney ER, Cave AE, Hohenberg MI. "We need a one-stop-shop": co-creating the model of care for a multidisciplinary memory clinic with community members, GPs, aged care workers, service providers, and policy-makers. BMC Geriatr. 2020 Feb 11;20(1):49. doi: 10.1186/s12877-019-1410-x. PMID 32046657
- [Background] Prince M, Bryce R, Albanese E, Wimo A, Ribeiro W, Ferri CP. The global prevalence of dementia: a systematic review and metaanalysis. Alzheimers Dement. 2013 Jan;9(1):63-75.e2. doi: 10.1016/j.jalz.2012.11.007. PMID 23305823
- [Background] Sachdev PS, Lipnicki DM, Kochan NA, Crawford JD, Thalamuthu A, Andrews G, Brayne C, Matthews FE, Stephan BC, Lipton RB, Katz MJ, Ritchie K, Carriere I, Ancelin ML, Lam LC, Wong CH, Fung AW, Guaita A, Vaccaro R, Davin A, Ganguli M, Dodge H, Hughes T, Anstey KJ, Cherbuin N, Butterworth P, Ng TP, Gao Q, Reppermund S, Brodaty H, Schupf N, Manly J, Stern Y, Lobo A, Lopez-Anton R, Santabarbara J; Cohort Studies of Memory in an International Consortium (COSMIC). The Prevalence of Mild Cognitive Impairment in Diverse Geographical and Ethnocultural Regions: The COSMIC Collaboration. PLoS One. 2015 Nov 5;10(11):e0142388. doi: 10.1371/journal.pone.0142388. eCollection 2015. PMID 26539987
- [Background] Bacigalupo I, Mayer F, Lacorte E, Di Pucchio A, Marzolini F, Canevelli M, Di Fiandra T, Vanacore N. A Systematic Review and Meta-Analysis on the Prevalence of Dementia in Europe: Estimates from the Highest-Quality Studies Adopting the DSM IV Diagnostic Criteria. J Alzheimers Dis. 2018;66(4):1471-1481. doi: 10.3233/JAD-180416. PMID 30412486
- See also: WHO (2021) Global Status report in the public health response to dementia — https://iris.who.int/bitstream/handle/10665/344701/9789240033245-eng.pdf?sequence=1
- See also: Istat 2024 — https://demo.istat.it/app/?i=POS&l=it
- See also: Gauthier S, Rosa-Neto P, Morais JA, & Webster C. (2021) World Alzheimer Report 2021, Abridged version: journey through the diagnosis of dementia. London, England: Alzheimer's Disease International. — https://www.alzint.org/u/World-Alzheimer-Report-2021.pdf